CLINICAL TRIAL: NCT00474487
Title: A Phase 3, Multi-center Study to Evaluate Safety and Immune Response of Novartis Meningococcal ACWY Conjugate Vaccine In Adults and Compare to the Safety and Immune Response of a Licensed Conjugate Meningococcal ACWY Vaccine in Subjects Aged 19-55 Years of Age and to a Licensed Polysaccharide Vaccine in Subjects Aged 56-65 Years of Age.
Brief Title: A Study to Evaluate Safety and Immune Response of Novartis Meningococcal ACWY Vaccine In Healthy Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V59P17
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2010-08-04 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-04

CONDITIONS: Meningococcal Meningitis; Meningococcal Infections
Keywords: Meningococcal; meningitis; vaccine; adolescents; adults
MeSH Terms: conditions — Meningitis, Meningococcal; Meningococcal Infections; Meningitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Novartis MenACWY Vaccine (19 to 55 Years) (Experimental): Novartis meningococcal ACWY conjugate vaccine administered to subjects 19 years to 55 years
  Interventions: Biological: MenACWY CRM (19 to 55 years)
- Licensed polysaccharide vaccine (Active Comparator): Licensed meningococcal ACWY polysaccharide vaccine
  Interventions: Biological: Meningococcal ACWY Polysaccharide Vaccine
- Licensed Conjugate Vaccine (Active Comparator): Licensed meningococcal ACWY polysaccharide-protein conjugate vaccine
  Interventions: Biological: Meningococcal ACWY Conjugate Vaccine
- Novartis MenACWY Vaccine (56 to 65 Years) (Experimental): Novartis meningococcal ACWY conjugate vaccine administered to subjects 56 years to 65 years
  Interventions: Biological: Novartis MenACWY Vaccine (56 to 65 Years)

INTERVENTIONS:
Biological: Meningococcal ACWY Polysaccharide Vaccine — One dose of the licensed meningococcal ACWY polysaccharide vaccine was administered by subcutaneous injection.
  Arms: Licensed polysaccharide vaccine
Biological: MenACWY CRM (19 to 55 years) — One dose of the Novartis meningococcal ACWY conjugate vaccine was administered by intramuscular injection to subjects 19 years to 55 years of age.
  Arms: Novartis MenACWY Vaccine (19 to 55 Years)
Biological: Meningococcal ACWY Conjugate Vaccine — One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered by intramuscular injection.
  Arms: Licensed Conjugate Vaccine
Biological: Novartis MenACWY Vaccine (56 to 65 Years) — One dose of the Novartis meningococcal ACWY conjugate vaccine was administered by intramuscular injection administered to subjects 56 years to 65 years of age.
  Arms: Novartis MenACWY Vaccine (56 to 65 Years)

SUMMARY:
This study will evaluate the safety and immune response of Novartis Meningococcal ACWY conjugate vaccine in healthy adolescents and adults.

ELIGIBILITY:
Inclusion Criteria:

* individuals who are 19-65 years of age inclusive and who, after the nature of the study has been explained have provided written informed consent
* individuals who are available for all visits and telephone calls scheduled for the study;
* individuals who are in good health

Exclusion Criteria:

* individuals with a previous or suspected disease caused by N. meningitidis
* individuals with previous immunization with a meningococcal vaccine or vaccine containing meningococcal antigen(s)
* individuals with previous or suspected disease caused by N. meningitidis
* individuals with any serious acute, chronic or progressive disease
* individuals who are pregnant or breastfeeding

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2831 (Actual)
Dates: Start 2007-05; Primary Completion 2007-08 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Director — Novartis
Locations (2):
- Buenos Aires, Argentina, Buenos Aires, Argentina
- Cali, Colombia; Bogota, Colombia, Cali; Bogota, Colombia

REFERENCES:
- [Result] Stamboulian D, Lopardo G, Lopez P, Cortes-Barbosa C, Valencia A, Bedell L, Karsten A, Dull PM. Safety and immunogenicity of an investigational quadrivalent meningococcal CRM(197) conjugate vaccine, MenACWY-CRM, compared with licensed vaccines in adults in Latin America. Int J Infect Dis. 2010 Oct;14(10):e868-75. doi: 10.1016/j.ijid.2010.03.017. Epub 2010 Jul 22. PMID 20655261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at 3 centers in Argentina and Colombia.
Pre-assignment Details: All subjects enrolled were included in the trial.
Groups:
- Novartis MenACWY Vaccine (19 to 55 Years); Novartis MenACWY Vaccine (56 to 65 Years): One dose (0.5 mL of injectable solution) of the Novartis meningococcal ACWY conjugate vaccine was administered intramuscularly after reconstitution.
- Licensed Conjugate Vaccine (19 to 55 Years): One 0.5 mL dose of the licensed meningococcal ACWY conjugate vaccine was administered intramuscularly (Ages 19 to 55 years).
- Licensed Polysaccharide Vaccine (56 to 65 Years): One 0.5 mL dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered subcutaneously(Ages 56 to 65 Years) after reconstitution.
Period: Overall Study
Arm/Group | Novartis MenACWY Vaccine (19 to 55 Years) | Novartis MenACWY Vaccine (56 to 65 Years) | Licensed Conjugate Vaccine (19 to 55 Years) | Licensed Polysaccharide Vaccine (56 to 65 Years)
Started | 1606 | 217 | 899 | 109
Completed | 1576 | 215 | 885 | 109
Not Completed | 30 | 2 | 14 | 0
Not completed — Withdrawal by Subject | 6 | 0 | 0 | 0
Not completed — Lost to Follow-up | 20 | 1 | 7 | 0
Not completed — Inappropriate enrollment | 4 | 0 | 7 | 0
Not completed — Death | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Novartis MenACWY Vaccine (19 to 55 Years) | Novartis MenACWY Vaccine (56 to 65 Years) | Licensed Conjugate Vaccine (19 to 55 Years) | Licensed Polysaccharide Vaccine (56 to 65 Years) | Total
Number analyzed (Participants) | 1606 | 217 | 899 | 109 | 2831
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.6 (10.1) | 60.1 (2.7) | 34.8 (10.4) | 60.1 (2.6) | 37.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1092 | 163 | 627 | 79 | 1961
  Male | 514 | 54 | 272 | 30 | 870
Race/Ethnicity, Customized [Number; unit: Subjects]
  Asian | 1 | 1 | 1 | 0 | 3
  Black | 135 | 18 | 109 | 8 | 270
  Caucasian | 249 | 38 | 127 | 23 | 437
  Hispanic | 1217 | 158 | 658 | 77 | 2110
  Other | 4 | 2 | 3 | 1 | 10
  Not Available | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least One Severe Systemic Reaction, Ages 19 to 55 Years
Description: Safety of the Novartis MenACWY conjugate vaccine and of a licensed meningococcal ACWY conjugate vaccine as measured by the number of subjects presenting at least one severe systemic reaction during the first 7 days following a single vaccination in healthy subjects.
Time Frame: Days 1 to 7
Population: The analysis was performed on the safety set. The number of subjects in the safety set is less than the randomized set due to premature withdrawals.
Measure: Number; unit: Subjects
Groups:
- Novartis MenACWY Vaccine: One dose of the Novartis meningococcal ACWY conjugate vaccine was administered intramuscularly.
- Licensed Conjugate Vaccine: One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Vaccine | Licensed Conjugate Vaccine
Number analyzed (Participants) | 1588 | 882
Subjects | 95 | 46

2. Secondary Outcome: Percentage of Subjects With Seroresponse and hSBA ≥ 1:8 (Ages 19 to 55 Years), PP Population
Description: Immunogenicity of the MenACWY vaccine and of a licensed meningococcal ACWY conjugate vaccine, defined as percentage of subjects with seroresponse, human Serum Bactericidal Activity (hSBA) ≥ 1:8 directed against N meningitidis serogroups A, C, W, and Y (healthy subjects aged 19 to 55 years).
  Seroresponse: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | Novartis MenACWY Vaccine | Licensed Conjugate Vaccine
Number analyzed (Participants) | 179 | 182
Percentage of subjects
  Seroresponders in serogroup A | 78 [71 to 84] | 77 [71 to 83]
  Seroresponders in serogroup C (N= 180, 183) | 83 [76 to 88] | 81 [74 to 86]
  Seroresponders in serogroup W (N= 178, 180) | 66 [58 to 73] | 53 [46 to 61]
  Seroresponders in serogroup Y (N= 181, 182) | 80 [74 to 86] | 58 [51 to 65]
  hSBA ≥1:8 in serogroup A | 81 [74 to 86] | 80 [74 to 86]
  hSBA ≥1:8 in serogroup C (N= 180, 183) | 88 [82 to 92] | 92 [87 to 96]
  hSBA ≥1:8 in serogroup W (N= 178, 180) | 98 [95 to 100] | 93 [89 to 97]
  hSBA ≥1:8 in serogroup Y (N= 181, 182) | 88 [82 to 92] | 76 [70 to 82]

3. Secondary Outcome: Percentage of Subjects With Seroresponse and hSBA ≥ 1:8 (Ages 56 to 65 Years), PP Population
Description: Immunogenicity of the MenACWY vaccine and of a licensed meningococcal ACWY conjugate vaccine, defined as percentage of subjects with seroresponse, human Serum Bactericidal Activity (hSBA) ≥ 1:8 directed against N meningitidis serogroups A, C, W, and Y (healthy subjects aged 56 to 65 years).
  Seroresponse: For a subject with hSBA titer <1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer ≥ 1:8; for a subject with hSBA titer ≥ 1:4 at baseline, seroresponse is defined as a postvaccination hSBA titer of at least 4 times the baseline.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Groups:
- Licensed Polysaccharide Vaccine: One dose of the licensed meningococcal ACWY polysaccharide vaccine administered subcutaneously.
Arm/Group | Novartis MenACWY Vaccine | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 83 | 41
Percentage of subjects
  Seroresponders in serogroup A | 86 [76 to 92] | 61 [45 to 76]
  Seroresponders in serogroup C (N= 84, 41) | 83 [74 to 91] | 73 [57 to 86]
  Seroresponders in serogroup W (N= 82, 39) | 61 [50 to 72] | 54 [37 to 70]
  Seroresponders in serogroup Y (N= 84, 41) | 77 [67 to 86] | 54 [37 to 69]
  hSBA ≥1:8 in serogroup A | 87 [78 to 93] | 63 [47 to 78]
  hSBA ≥1:8 in serogroup C (N= 84, 41) | 90 [82 to 96] | 83 [68 to 93]
  hSBA ≥1:8 in serogroup W (N= 82, 39) | 94 [86 to 98] | 95 [83 to 99]
  hSBA ≥1:8 in serogroup Y (N= 84, 41) | 88 [79 to 94] | 68 [52 to 82]

4. Secondary Outcome: Summary of hSBA GMTs (Ages 19 to 55 Years), PP Population
Description: Immunogenicity of a single dose of MenACWY and of a single dose of the licensed meningococcal ACWY conjugate vaccine, as measured by serum bactericidal activity geometric mean titer (GMT) response using human complement (hSBA GMTs) directed against N meningitidis serogroups A, C, W-135, and Y at 1 month after vaccination, when administered to healthy subjects 19 to 55 years of age.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Novartis MenACWY Vaccine | Licensed Conjugate Vaccine
Number analyzed (Participants) | 179 | 182
Titers
  Serogroup A | 77 [57 to 105] | 52 [38 to 70]
  Serogroup C (N=180, 183) | 114 [84 to 153] | 88 [65 to 118]
  Serogroup W (N=178, 180) | 159 [123 to 205] | 112 [87 to 144]
  Serogroup Y (N=181, 182) | 95 [70 to 127] | 40 [30 to 54]

5. Secondary Outcome: Summary of hSBA GMTs (Ages 56 to 65 Years), PP Population
Description: Immunogenicity of a single dose of MenACWY and of a single dose of the licensed meningococcal ACWY conjugate vaccine, as measured by serum bactericidal activity geometric mean titer (GMT) response using human complement (hSBA GMTs) directed against N meningitidis serogroups A, C, W-135, and Y at 1 month after vaccination, when administered to healthy subjects 56 to 65 years of age.
Time Frame: 1 month postvaccination
Population: The analysis was performed on the per-protocol (PP) population.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Novartis MenACWY Vaccine | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 83 | 41
Titers
  Serogroup A | 111 [70 to 175] | 21 [11 to 39]
  Serogroup C (N=84, 41) | 196 [125 to 306] | 86 [45 to 163]
  Serogroup W (N=82, 39) | 164 [112 to 240] | 132 [76 to 229]
  Serogroup Y (N=84, 41) | 121 [76 to 193] | 28 [15 to 55]

6. Secondary Outcome: Number of Subjects With Local and Systemic Reactions, Ages 19 to 55 Years
Description: Safety profile following a single vaccination of MenACWY CRM vaccine and of a single vaccination of a licensed meningococcal ACWY conjugate vaccine administered to healthy subjects (ages 19 to 55 years).
Time Frame: Days 1 to 7
Population: The analysis was performed on the safety population.
Measure: Number; unit: Subjects
Arm/Group | Novartis MenACWY Vaccine | Licensed Conjugate Vaccine
Number analyzed (Participants) | 1588 | 882
Subjects
  Any local reaction | 729 | 439
  Pain | 632 | 392
  Erythema | 207 | 105
  Induration | 179 | 115
  Any systemic reaction | 616 | 375
  Chills | 124 | 70
  Nausea | 112 | 77
  Malaise | 309 | 186
  Myalgia | 197 | 131
  Arthralgia | 118 | 76
  Headache | 421 | 254
  Rash | 53 | 22
  Fever ≥38°C (N= 1587, 882) | 56 | 31
  Any Other Reaction | 280 | 162
  Analgesic/Antipyretic Med. Used (N=1588, 881) | 250 | 148
  Stayed Home (N= 1585, 880) | 75 | 46

7. Secondary Outcome: Number of Subjects With Local and Systemic Reactions, Ages 56 to 65 Years
Description: Safety profile following a single vaccination of MenACWY vaccine and of a single vaccination of a licensed meninococcal ACWY polysaccharide vaccine administered to healthy subjects (ages 56 to 65 years).
Time Frame: Days 1 to 7
Population: The analysis was done on the safety population.
Measure: Number; unit: Subjects
Groups:
- Licensed Polysaccharide Vaccine: One dose of the licensed meningococcal ACWY polysaccharide vaccine was administered intramuscularly.
Arm/Group | Novartis MenACWY Vaccine | Licensed Polysaccharide Vaccine
Number analyzed (Participants) | 216 | 109
Subjects
  Any local reaction | 92 | 44
  Pain | 69 | 34
  Erythema | 41 | 13
  Induration | 39 | 17
  Any systemic reaction | 84 | 44
  Chills | 26 | 6
  Nausea | 20 | 8
  Malaise | 50 | 20
  Myalgia | 39 | 11
  Arthralgia | 25 | 11
  Headache | 52 | 30
  Rash | 10 | 2
  Fever ≥38°C | 6 | 3
  Any other reaction | 29 | 15
  Analgesic/Antipyretic Med. Used | 25 | 14
  Stayed Home (N= 214, 108) | 14 | 6

ADVERSE EVENTS:
Time Frame: Serious adverse events were collected from study day 1 to 180.
Description: The analysis was performed on the safety set. The number of subjects in the safety set is less than the randomized set due to premature withdrawals.
Groups:
- Novartis MenACWY Vaccine (19 to 55 Years); Novartis MenACWY Vaccine (56 to 65 Years): One dose of the Novartis meningococcal ACWY conjugate vaccine was administered intramuscularly.
- Licensed Conjugate Vaccine (19 to 55 Years): One dose of the licensed meningococcal ACWY polysaccharide-protein conjugate vaccine was administered intramuscularly in ages 19 to 55 years.
- Licensed Polysaccharide Vaccine (56 to 65 Years): One dose of the licensed meningococcal ACWY polysaccharide vaccine was administered intramuscularly (Ages 56 to 65 Years)
Arm/Group | Novartis MenACWY Vaccine (19 to 55 Years) | Novartis MenACWY Vaccine (56 to 65 Years) | Licensed Conjugate Vaccine (19 to 55 Years) | Licensed Polysaccharide Vaccine (56 to 65 Years)
Serious Adverse Events (participants affected / at risk) | 11/1588 | 1/216 | 8/882 | 1/109
Other Adverse Events (participants affected / at risk) | 955/1588 | 124/216 | 561/882 | 62/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novartis MenACWY Vaccine (19 to 55 Years) (N=1588) | Novartis MenACWY Vaccine (56 to 65 Years) (N=216) | Licensed Conjugate Vaccine (19 to 55 Years) (N=882) | Licensed Polysaccharide Vaccine (56 to 65 Years) (N=109)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Generalised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIV Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pelvic Inflammatory disease (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyometra (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthropod Sting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Limb Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nephrectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypovolaemic Shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Novartis MenACWY Vaccine (19 to 55 Years) (N=1588) | Novartis MenACWY Vaccine (56 to 65 Years) (N=216) | Licensed Conjugate Vaccine (19 to 55 Years) (N=882) | Licensed Polysaccharide Vaccine (56 to 65 Years) (N=109)
Injection site pain (General disorders) | 632 | 69 | 392 | 34
Injection site erythema (General disorders) | 207 | 41 | 105 | 13
Injection site induration (General disorders) | 179 | 39 | 115 | 17 — N= 1588, 216, 882, 108
Chills (General disorders) | 124 | 26 | 70 | 6
Nausea (Gastrointestinal disorders) | 112 | 20 | 77 | 8
Malaise (General disorders) | 309 | 50 | 186 | 20
Myalgia (Musculoskeletal and connective tissue disorders) | 197 | 39 | 131 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 118 | 25 | 76 | 11
Headache (Nervous system disorders) | 421 | 52 | 254 | 30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No